CLINICAL TRIAL: NCT04645407
Title: Efficacy of Fuzheng Huayu Tablets for Treating Pulmonary Inflammation in Patients With COVID-19: A Case-Control Study
Brief Title: Effects of Fuzheng Huayu Tablets on COVID-19
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ShuGuang Hospital (Other)
Collaborators: Hubei Hospital of Traditional Chinese Medicine (Other); Jingmen No.1 People's Hospital (Other)
Responsible Party: Principal Investigator, Liu Chenghai, Institute Director;PhD, ShuGuang Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Fzhy-ncp-1
Record Dates: First submitted 2020-02-15; First posted 2020-11-27 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Novel Coronavirus Pneumonia
MeSH Terms: interventions — fuzheng huayu

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FZHY Group (Experimental): conventional therapy plus Fuzheng Huayu tablet (0.4g/tablet, 1.6g/time, 3 times/day, oral; take medicine after meals each time.)
  Interventions: Drug: Fuzheng Huayu tablet
- Control Group (No Intervention): conventional therapy

INTERVENTIONS:
Drug: Fuzheng Huayu tablet — Fuzheng Huayu tablet (0.4g/tablet, 1.6g/time, 3 times/day, oral; take medicine after meals each time)
  Arms: FZHY Group

SUMMARY:
The 2019 novel coronavirus (2019-nCoV) infection caused clusters of severe respiratory illness similar to SARS and was associated with ICU admission and high mortality. There is no confirmed antivirus therapy for people infected 2019-nCoV, most of them should receive supportive care to help relieve symptoms. This clinical trial is to evaluate the effect of Fuzheng Huayu tablet on lung inflammation in intensive patients with novel coronavirus pneumonia and reduce the progressive rate to critical type.

DETAILED DESCRIPTION:
In December 2019, new coronavirus pneumonia (NCP) occurred in Wuhan, Hubei Province, which spread rapidly. Some of the patients developed into severe or critical illness. It became an international concerned public health emergencies and one of the major epidemics seriously endangering people's health and public safety after severe acute respiratory syndrome (SARS) in 2003.

At present, we lack the specific treatment for NCP. The anti- novel coronavirus drugs are been conducting in clinical trials, and the other options includes the symptomatic treatment. The pathological mechanism of the disease is not clear, but due to the continuous development of inflammation, some cases can become severe or critical, which threatening the life and health of patients. Intensive cases with obvious inflammation, after the control of acute symptoms and signs, often have the performance of pulmonary fibrosis, affecting the recovery of lung function. Therefore, actively reducing lung inflammation, controlling and reversing pulmonary fibrosis is of great significance for the life and health of patients Infected novel coronavirus.

Our previous study found that Fuzheng Huayu prescription can reduce the inflammation and fibrosis of the lung in the model rats, and improve the lung function of the patients with COPD. Therefore, we hope to take Fuzheng Huayu tablet to NCP patients, and observe whether it can reduce the lung inflammation of patients, so as to reduce the rate of progression of critical illness.

ELIGIBILITY:
Inclusion Criteria:

Patients were included if they (1) had COVID-19; (2) were 18 to 65 years old; (3) did not participate in other drug clinical studies within 1 month before enrollment; and (4) voluntarily accepted treatment and signed an informed consent form.

Exclusion Criteria:

Patients were excluded if they (1) had critical COVID-19; (2) were unconsciousness, had dementia, had psychiatric conditions, or were unable to communicate normally; (3) had severe cardiac insufficiency (i.e., cardiac function grade IV), severe liver or kidney disease, bronchial asthma, COPD, neurological disease, tumor, thoracic deformity, or immunodeficiency disease; (4) were pregnant or lactating or had a recent pregnancy plan; and (5) had a known allergy to any treatment drug.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-04-15 (Actual)

PRIMARY OUTCOMES:
the percentage of patients showing improvement in chest CT | Week 2
  Evaluation of the therapeutic effect of Fuzheng huayu tablet

SECONDARY OUTCOMES:
remission rate or progression rate of critical illness | Week 2
  Evaluation of pulmonary inflammation improvement
clinical remission rate of respiratory symptoms | week 2
  Evaluation of pulmonary inflammation improvement
routine blood examination | Week 2
  Evaluation of pulmonary inflammation improvement
C-reactive protein level | Week 2
  Evaluation of the therapeutic effect of Fuzheng huayu tablet
procalcitonin level | Week 2
  Evaluation of pulmonary inflammation improvement
oxygen saturation | Week 2
  Evaluation of pulmonary inflammation improvement

CONTACTS AND LOCATIONS:
Locations (1):
- Shuguang Hospital, Shanghai, Shanghai Municipality, China